CLINICAL TRIAL: NCT01100606
Title: A Multicenter, Randomized, Open-Label, Crossover Study to Evaluate the Mode of Administration and Safety of EUR-1008 in Infants 1 to 12 Months of Age With Exocrine Pancreatic Insufficiency (EPI) Associated With Cystic Fibrosis (CF)
Brief Title: A Study to Evaluate the Mode of Administration and Safety of EUR-1008 (APT-1008) in Infants 1 to 12 Months of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PR-011
Record Dates: First submitted 2010-03-31; First posted 2010-04-09 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-03

CONDITIONS: Cystic Fibrosis; Exocrine Pancreatic Insufficiency
Keywords: Exocrine Pancreatic Insufficiency; Infants with CF
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUR-1008 (APT-1008) in Apple Juice (Experimental)
  Interventions: Drug: EUR-1008 (APT-1008)
- EUR-1008 (APT-1008) in Apple Sauce (Experimental)
  Interventions: Drug: EUR-1008 (APT-1008)

INTERVENTIONS:
Drug: EUR-1008 (APT-1008) — EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) from open capsule, mixed with a small amount of apple juice, will be given orally daily using a syringe nurser at dose increments of 3,000 lipase units, for 10 days in either first treatment period or second treatment period. Total dose will not exceed 10,000 lipase units per kilogram (kg) of body weight per day.
  Other Names: Zenpep® (pancrelipase) delayed release capsules
  Arms: EUR-1008 (APT-1008) in Apple Juice
Drug: EUR-1008 (APT-1008) — EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) from open capsule, mixed with a small amount of apple sauce, will be given orally daily using a spoon at dose increments of 3,000 lipase units, for 10 days in either first treatment period or second treatment period. Total dose will not exceed 10,000 lipase units per kg of body weight per day.
  Other Names: Zenpep® (pancrelipase) delayed release capsules
  Arms: EUR-1008 (APT-1008) in Apple Sauce

SUMMARY:
A study to determine the safety, effectiveness, and acceptability of 2 methods of administration of EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) 3,000 lipase units capsule, a pancreatic enzyme product (PEP), in infants with exocrine pancreatic insufficiency (EPI) due to cystic fibrosis (CF). This study is sponsored by Aptalis Pharma (formerly Eurand).

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, crossover study in pediatric participants with EPI due to CF. The study will be carried out in infants between 1 and 12 months of age.

The study comprises of a screening period (up to 10 days) followed by 2 treatment periods (10 days each). During the screening period, all participants will be administered Zenpep® 5,000 (pancrelipase) mixed with a small amount of apple sauce. Once determined eligible for participation, participants will be randomized into 1 of 2 treatment sequences. Each sequence corresponds to taking one treatment in the first period and the other treatment in the second period, and were administered EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) 3,000 lipase units capsule either mixed with apple juice using a syringe nurser or apple sauce using a spoon.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of CF based on the following criteria: one clinical feature consistent with CF, and either a genotype with 2 identifiable mutations known to cause CF or a sweat chloride concentration that is greater than 60 milliequivalent per liter by quantitative pilocarpine iontophoresis
* Participants who have the need for a PEP defined as monoclonal fecal elastase less than 200 microgram per gram (mcg/g) stool
* Caregiver must be willing to switch participant from their previous PEP (if any) to Zenpep®
* Participants who have a height to weight ratio target at greater than tenth percentile
* Participants who are clinically stable with no evidence of concomitant illness or acute upper or lower respiratory tract infection during the 7-day interval prior to screening and preceding accession into this clinical study

Exclusion Criteria:

* Participants who are less than 1 month old or are greater than 12 months old
* Participants with history of meconium ileus or small bowel atresia in the newborn period that required surgery
* Participants who are allergic to pork or other porcine PEPs
* Participants with any respiratory condition or other serious comorbidity (for example patent ductus arteriosus [PDA], or necrotizing enterocolitis [NEC]) that in the investigator's opinion would result in an intervention requiring hospitalization or intensive pulmonary or other treatment during the trial
* Participants with other comorbidities independent of CF that, in the investigator's opinion, would result in an inability to participate in the study or excess risk to the participant that is above the standard of care
* Participants with acute respiratory infection in the previous 14 days requiring antibiotics
* Participants who required change in antacid dose in the 7 days before screening
* Participants with administration of oral, intramuscular (IM), intravenous (IV) glucocorticoids in the 4 weeks prior to screening
* Participants with any condition that would, in the investigator's opinion, limit the participant's ability to complete the study
* Participants currently participating in or has participated in an investigational study, with the exception of observational studies, within 30 days of the screening visit

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (6):
- United States (6):
  - Nemours Children's Clinic, Jacksonville, Florida
  - Children's Lung Specialists Ltd., Las Vegas, Nevada
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Cystic Fibrosis Care Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants were administered Zenpep® 5,000 (pancrelipase) from open capsule mixed with a small amount of apple sauce in the screening period for 10 days.
Groups:
- EUR-1008 (APT-1008) in Apple Juice First, Then in Apple Sauce: EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) from open capsule, mixed with a small amount of apple juice using a syringe nurser, orally daily at dose increments of 3,000 lipase units, for 10 days in first treatment period followed by EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) from open capsule, mixed with a small amount of apple sauce using a spoon, orally daily at dose increments of 3,000 lipase units, for 10 days in second treatment period. Total dose was not to exceed 10,000 lipase units/kilogram body weight/day (lipase units/kg/day).
- EUR-1008 (APT-1008) in Apple Sauce First, Then in Apple Juice: EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) from open capsule, mixed with a small amount of apple sauce using a spoon, orally daily at dose increments of 3,000 lipase units, for 10 days in first treatment period followed by EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) from open capsule, mixed with a small amount of apple juice using a syringe nurser, orally daily at dose increments of 3,000 lipase units, for 10 days in second treatment period. Total dose was not to exceed 10,000 lipase units/kg/day.
Period: First Treatment Period
Arm/Group | EUR-1008 (APT-1008) in Apple Juice First, Then in Apple Sauce | EUR-1008 (APT-1008) in Apple Sauce First, Then in Apple Juice
Started | 8 | 7
Completed | 8 (Due to difficulty with syringe nurser,1 participant completed study with apple sauce,not apple juice) | 7
Not Completed | 0 | 0
Period: Second Treatment Period
Arm/Group | EUR-1008 (APT-1008) in Apple Juice First, Then in Apple Sauce | EUR-1008 (APT-1008) in Apple Sauce First, Then in Apple Juice
Started | 8 | 7
Completed | 8 (Due to intolerance to apple sauce & apple juice,1 participant completed study with banana-based food) | 7 (Due to difficulty with syringe nurser, 1 participant completed study using apple sauce)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of study medication.
Groups:
- Entire Study Population: Includes all enrolled participants who received EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) mixed with a small amount of apple juice using a syringe nurser first and EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) mixed with a small amount of apple sauce using a spoon first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.7 (3.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Average Daily Number of Stools [Mean (Standard Deviation); unit: average number of stools per day] — Average daily number of stools of each participant was calculated from frequency of stools by the participant per day. Average daily number of stools during the screening period for total participants was summarized. Number of participants evaluable for this baseline characteristic was 12.
  average number of stools per day | 2.73 (1.393)
Number of Stools Categorized as Per Consistency [Mean (Standard Deviation); unit: average number of stools per day] — Stool consistency was categorized as hard, formed/normal, soft and diarrhea. Average number of stools categorized as per consistency of each participant was calculated from number of stools of specific consistency by the participant per day. Average number of stools categorized as per consistency during the screening period for total participants was summarized. Number of participants evaluable for this baseline characteristic was 12.
  average number of stools per day
    Hard | 0.11 (0.255)
    Normal | 1.18 (1.129)
    Soft | 0.91 (0.777)
    Diarrhea | 0.48 (0.801)
Number of Stools With Signs of Blood and Visible Oil or Grease [Mean (Standard Deviation); unit: average number of stools per day] — Average number of stools with signs of blood and visible oil or grease of each participant was calculated from number of stools with signs of blood and visible oil or grease by the participant per day. Average number of stools stools with signs of blood and visible oil or grease during the screening period for total participants was summarized. Number of participants evaluable for this baseline characteristic was 12.
  average number of stools per day
    With blood | 0 (0)
    With visible oil or grease | 0.11 (0.147)
Number of Abdominal Symptoms: Bloating [Mean (Standard Deviation); unit: average number of bloating per day] — Bloating is swelling of the intestinal tract caused by excessive gas formation. Symptoms of bloating were classified by severity as 0=none, 1=mild (no impairment of daily activities), 2=moderate (slight impairment of daily activities), and 3=severe (unable to perform daily activities). Average number of symptoms of specific severity for each participant was calculated from frequency of symptoms by the participant per day. Average number of symptoms during the screening period for total participants was summarized. Number of participants evaluable for this baseline characteristic was 12.
  average number of bloating per day
    Mild Bloating | 0.12 (0.281)
    Moderate Bloating | 0.04 (0.101)
    Severe Bloating | 0 (0)
Number of Abdominal Symptoms: Flatulence [Mean (Standard Deviation); unit: average number of flatulence per day] — Flatulence is presence of excessive gas in the digestive tract. Symptoms of flatulence were classified by severity as 0=none, 1=mild (no impairment of daily activities), 2=moderate (slight impairment of daily activities), and 3=severe (unable to perform daily activities). Average number of symptoms of specific severity for each participant was calculated from frequency of symptoms by the participant per day. Average number of symptoms during the screening period for total participants was summarized. Number of participants evaluable for this baseline characteristic was 12.
  average number of flatulence per day
    Mild Flatulence | 1.00 (1.208)
    Moderate Flatulence | 0.51 (0.728)
    Severe Flatulence | 0.03 (0.099)
Number of Abdominal Pain Symptoms [Mean (Standard Deviation); unit: average number of pain symptoms per day] — Symptoms of pain was classified by severity as 0=none, 1=mild (no impairment of daily activities), 2=moderate (slight impairment of daily activities), and 3=severe (unable to perform daily activities). Average number of symptoms of specific severity for each participant was calculated from frequency of symptoms by the participant per day. Average number of symptoms during the screening period for total participants was summarized. Number of participants evaluable for this baseline characteristic was 12.
  average number of pain symptoms per day
    Mild Abdominal Pain | 0.23 (0.409)
    Moderate Abdominal Pain | 0.09 (0.185)
    Severe Abdominal Pain | 0.02 (0.066)

OUTCOME MEASURES:

1. Secondary Outcome: Daily Number of Stools
Description: Average daily number of stools of each participant was calculated from frequency of stools by the participant per day. Average daily number of stools during the first treatment period, second treatment period and end of study for total participants was summarized.
Time Frame: Up to Day 10 in first and second treatment periods, end of study (Day 21)
Population: ITT population included all participants who received at least 1 dose of study medication, had data (partial or complete) on acceptability questionnaire on and clinical signs and symptoms of EPI. Here, 'N' (number of participants analyzed) =participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: average number of stools per day
Groups:
- EUR-1008 (APT-1008) in Apple Juice: EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) from open capsule, mixed with a small amount of apple juice using a syringe nurser, orally daily at dose increments of 3,000 lipase units, for 10 days in either first treatment period or second treatment period.
- EUR-1008 (APT-1008) in Apple Sauce: EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsule) from open capsule, mixed with a small amount of apple sauce using a spoon, orally daily at dose increments of 3,000 lipase units, for 10 days in either first treatment period or second treatment period.
Arm/Group | EUR-1008 (APT-1008) in Apple Juice | EUR-1008 (APT-1008) in Apple Sauce
Number analyzed (Participants) | 12 | 12
average number of stools per day | 2.76 (0.771) | 2.44 (0.766)

2. Secondary Outcome: Number of Stools Categorized as Per Consistency
Description: Stool consistency was categorized as hard, formed/normal, soft and diarrhea. Average number of stools categorized as per consistency of each participant was calculated from number of stools of specific consistency by the participant per day. Average number of stools categorized as per consistency during the first treatment period, second treatment period and end of study for total participants was summarized.
Time Frame: Up to Day 10 in first and second treatment periods, end of study (Day 21)
Population: ITT population included all participants who received at least 1 dose of study medication, had data (partial or complete) on acceptability questionnaire and clinical signs and symptoms of EPI. Here, 'N' (number of participants analyzed) =participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: average number of stools per day
Arm/Group | EUR-1008 (APT-1008) in Apple Juice | EUR-1008 (APT-1008) in Apple Sauce
Number analyzed (Participants) | 12 | 12
average number of stools per day
  Hard | 0.04 (0.089) | 0.14 (0.184)
  Normal | 1.77 (0.864) | 1.37 (0.770)
  Soft | 0.62 (0.710) | 0.83 (0.813)
  Diarrhea | 0.24 (0.527) | 0.07 (0.135)

3. Secondary Outcome: Number of Stools With Signs of Blood and Visible Oil or Grease
Description: Average number of stools with signs of blood and visible oil or grease of each participant was calculated from number of stools with signs of blood and visible oil or grease by the participant per day. Average number of stools with signs of blood and visible oil or grease during the first treatment period, second treatment period and end of study for total participants was summarized.
Time Frame: Up to Day 10 in first and second treatment periods, end of study (Day 21)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: average number of stools per day
Arm/Group | EUR-1008 (APT-1008) in Apple Juice | EUR-1008 (APT-1008) in Apple Sauce
Number analyzed (Participants) | 12 | 12
average number of stools per day
  With blood | 0 (0) | 0.01 (0.047)
  With visible oil or grease | 0.09 (0.191) | 0.17 (0.368)

4. Secondary Outcome: Number of Abdominal Symptoms: Bloating
Description: Bloating is swelling of the intestinal tract caused by excessive gas formation. Symptoms of bloating were classified by severity as 0=none, 1=mild (no impairment of daily activities), 2=moderate (slight impairment of daily activities), and 3=severe (unable to perform daily activities). Average number of symptoms of specific severity for each participant was calculated from frequency of symptoms by the participant per day. Average number of symptoms during the first treatment period, second treatment period and end of study for total participants was summarized.
Time Frame: Up to Day 10 in first and second treatment periods, end of study (Day 21)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: average number of bloating per day
Arm/Group | EUR-1008 (APT-1008) in Apple Juice | EUR-1008 (APT-1008) in Apple Sauce
Number analyzed (Participants) | 12 | 12
average number of bloating per day
  Mild Bloating | 0.22 (0.632) | 0.26 (0.857)
  Moderate Bloating | 0 (0) | 0 (0)
  Severe Bloating | 0 (0) | 0 (0)

5. Secondary Outcome: Number of Abdominal Symptoms: Flatulence
Description: Flatulence is presence of excessive gas in the digestive tract. Symptoms of flatulence were classified by severity as 0=none, 1=mild (no impairment of daily activities), 2=moderate (slight impairment of daily activities), and 3=severe (unable to perform daily activities). Average number of symptoms of specific severity for each participant was calculated from frequency of symptoms by the participant per day. Average number of symptoms during the first treatment period, second treatment period and end of study for total participants was summarized.
Time Frame: Up to Day 10 in first and second treatment periods, end of study (Day 21)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: average number of flatulence per day
Arm/Group | EUR-1008 (APT-1008) in Apple Juice | EUR-1008 (APT-1008) in Apple Sauce
Number analyzed (Participants) | 12 | 12
average number of flatulence per day
  Mild Flatulence | 1.0 (1.583) | 0.62 (0.869)
  Moderate Flatulence | 0.31 (0.559) | 0.32 (0.670)
  Severe Flatulence | 0.04 (0.144) | 0 (0)

6. Secondary Outcome: Number of Abdominal Pain Symptoms
Description: Symptoms of pain was classified by severity as 0=none, 1=mild (no impairment of daily activities), 2=moderate (slight impairment of daily activities), and 3=severe (unable to perform daily activities). Average number of symptoms of specific severity for each participant was calculated from frequency of symptoms by the participant per day. Average number of symptoms during the first treatment period, second treatment period and end of study for total participants was summarized.
Time Frame: Up to Day 10 in first and second treatment periods, end of study (Day 21)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: average number of pain symptoms per day
Arm/Group | EUR-1008 (APT-1008) in Apple Juice | EUR-1008 (APT-1008) in Apple Sauce
Number analyzed (Participants) | 12 | 12
average number of pain symptoms per day
  Mild Abdominal Pain | 0.10 (0.259) | 0.13 (0.343)
  Moderate Abdominal Pain | 0.09 (0.238) | 0.07 (0.231)
  Severe Abdominal Pain | 0 (0) | 0 (0)

7. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory and Vital Signs Findings
Time Frame: Baseline up to end of study (Day 21)
Population: Data was reported in individual participant listings but not statistically summarized for analysis as planned.
Arm/Group | EUR-1008 (APT-1008) in Apple Juice | EUR-1008 (APT-1008) in Apple Sauce
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormal Findings With Respect to Oral Mucosa
Description: Safety assessed by the presence of lesions observed during a physical examination at each visit. Severity of lesions measured by investigator's assessment using the following scale: mild = asymptomatic or mild symptoms and treatment not indicated; moderate = moderate pain but not interfering with oral intake, modified diet indicated; severe = severe pain, interfering with oral intake and life threatening or fatal.
Time Frame: Baseline up to end of study (Day 21)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | EUR-1008 (APT-1008) in Apple Juice | EUR-1008 (APT-1008) in Apple Sauce
Number analyzed (Participants) | 12 | 15
participants | 0 | 0

9. Primary Outcome: Treatment Difference for Acceptability of Treatment
Description: Acceptability questionnaire consists of 9 question (Q) to assess ease, time, overall satisfaction of study drug. Rated on 5-point scale for Q1-Q5 and Q7-Q9; Q6 was not rated and asked for name of previous PEP administered. Q1=overall ease of administration (1=not at all easy,2=somewhat,3=easy,4=very,5=extremely); Q2=time of administration (1=very short[<2 min],2=short[2-5 min],3=moderate[5-15 min],4=long[15-25 min],5=very long[>25 min]);Q3=overall infant acceptance(1=very easily,2=easily,3=same,4=with difficulty,5=with great difficulty);Q4=clear/complete instructions(1=not clear,2=somewhat,3=clear,4=very,5=extremely);Q5=overall satisfaction with dosing method (1=not satisfied,2=somewhat,3=satisfied,4=very,5=extremely);Q7=comparative ease of administration (1=much worse,2=worse,3=same,4=better,5=much better);Q8=comparative infant acceptance (1=much more difficult,2=more,3=same,4=easier,5=much easier);Q9=comparative overall satisfaction (1=much less,2=less,3=same,4=more,5=much more).
Time Frame: Baseline up to end of study (Day 21)
Population: Intention-to-treat (ITT) population included all participants who received at least 1 dose of study medication, had data (partial or complete) on acceptability questionnaire and clinical signs and symptoms of exocrine pancreatic insufficiency (EPI). Here, 'N' (number of participants analyzed) =participants who were evaluable for this measure.
Measure: Median (Full Range); unit: units on a scale
Groups:
- EUR-1008 (APT-1008) in Apple Juice: EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsules) from open capsule, mixed with a small amount of apple juice using a syringe nurser, orally daily with dose increments of 3,000 lipase units, for 10 days in either first treatment period or second treatment period.
- EUR-1008 (APT-1008) in Apple Sauce: EUR-1008 (APT-1008) (Zenpep® [pancrelipase] delayed release capsules) from open capsule, mixed with a small amount of apple sauce using a spoon, orally daily with dose increments of 3,000 lipase units, for 10 days in either first treatment period or second treatment period.
Arm/Group | EUR-1008 (APT-1008) in Apple Juice | EUR-1008 (APT-1008) in Apple Sauce
Number analyzed (Participants) | 12 | 12
units on a scale
  Ease of Administration | 1.5 [1 to 3] | 3.5 [2 to 5]
  Time of Administration | 2.5 [1 to 4] | 1.0 [1 to 3]
  Overall Infant Acceptance | 3.5 [2 to 5] | 1.5 [1 to 4]
  Dispensing Instructions | 3.0 [1 to 5] | 4.5 [3 to 5]
  Overall Satisfaction | 1.0 [1 to 3] | 3.0 [2 to 4]
  Comparative Ease of Administration | 2.0 [1 to 5] | 3.0 [2 to 5]
  Comparative Infant Acceptance | 2.0 [1 to 5] | 3.0 [3 to 5]
  Comparative Overall Satisfaction | 1.0 [1 to 4] | 3.0 [3 to 5]

10. Primary Outcome: Question 6 (Previous Pancreatic Enzyme Product [PEP])
Description: Acceptability questionnaire consists of 9 questions (Q) to assess the ease, time, overall satisfaction of study drug. Q6 included "name of previous PEP administered". Q6 was reported as number of participants who used any PEP prior to screening.
Time Frame: Baseline
Population: Safety analysis population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 15
participants
  Zenpep® | 4
  Creon® | 9
  Ultrase® | 1
  Pancrecarb® | 1

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (Day 21)
Description: Adverse event (AE): any untoward medical occurrence regardless of causal relationship to study drug. Serious AE: any event resulting in death, life threatening, required or prolonged in-patient hospitalization, significant disability/incapacity, or was congenital anomaly/birth defect. Participants at risk in EUR-1008 (APT-1008) in Apple Juice: 12
Groups:
- Zenpep®: Zenpep® 5,000 from open capsule, mixed with a small amount of apple sauce, orally daily in the screening period for 10 days.
Arm/Group | Zenpep® | EUR-1008 (APT-1008) in Apple Juice | EUR-1008 (APT-1008) in Apple Sauce
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 10/12 | 14/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zenpep® (N=15) | EUR-1008 (APT-1008) in Apple Juice (N=12) | EUR-1008 (APT-1008) in Apple Sauce (N=15)
Flatulence (Gastrointestinal disorders) | 6 | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1
Steatorrhoea (Gastrointestinal disorders) | 3 | 2 | 4
Teething (Gastrointestinal disorders) | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pyrexia (General disorders) | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Infantile spitting up (Gastrointestinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Drooling (Nervous system disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions vary in accordance with each agreement with the individual investigators. Sponsor will allow publication after a multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and can defer publication for a period of time to allow for Sponsor to obtain patent or other intellectual property right protection.